CLINICAL TRIAL: NCT05453461
Title: ADVANCED FSHD-COM: New Clinical Outcome Measures to Evaluate Non-ambulant FSHD Patients, a Pilot Study
Acronym: ADVANCED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-PP-06
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- new COMs for non ambulant FSHD patients (Experimental)
  Interventions: Diagnostic Test: Validation of new COMs for non ambulant FSHD patients

INTERVENTIONS:
Diagnostic Test: Validation of new COMs for non ambulant FSHD patients — Monitoring of commonly used and news COMs in non ambulant patients with facioscapulohumeral muscular dystrophy

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSHD) is one of the most common adult muscular dystrophy with an estimated prevalence range of 2-7 per 100,000. The disease is characterized by slowly progressive, asymmetric muscle weakness that starts with the face and scapular muscles. It causes significant lifetime morbidity, with up to 20% of patients eventually requiring full-time wheelchair use. However, there is a large degree of clinical variability in both disease progression and severity. This makes predicting an individual's disease course difficult and has made clinical trial design challenging.

The disease is caused by the aberrant expression of a normally silenced gene, DUX4, which causes disease by a toxic gain-of-function. The establishment of a unifying model for the cause of FSHD made it possible to develop disease-specific targeted treatments. Pharmaceutical companies are actively investigating therapeutic approaches in order to knockdown or silence DUX4, including the use of antisense RNA oligonucleotides which is already investigated for spinal muscular atrophy, Duchenne muscular dystrophy, and myotonic dystrophy. The drug development pipeline for FSHD over the next 5 years looks promising but meetings with industry, advocacy groups, and FSHD scientific experts have identified several gaps that need to be addressed to accelerate efficient drug development. As drugs move from preclinical testing into human trials, it is essential to validate clinical trial tools and methodologies to facilitate drug development. There is a strong need for clinical outcome measures (COMs) including biomarkers, strength outcomes, functional measures and patient reported outcomes to follow disease progression and to evaluate treatment efficacy.

A large international multicenter study is currently ongoing in order to validate COMs in ambulant FSHD patients (ReSolve, NCT03458832). Additionally, Nice University Hospital is conducting an ancillary study (CTRL FSHD France, NCT04038138) to evaluate muscle MRI, an additional emerging biomarker, to follow disease progression in the same patient population. To limit patient heterogeneity, only ambulant FSHD patients are included in these 2 ongoing studies. It is therefore important to generate data in severely affected non-ambulant FSHD patients, in order to validate COMs that are adapted to this specific subgroup of patients for future therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed FSHD1 or clinical diagnosis of FSHD with characteristic findings on exam and an affected parent or offspring
* Age 18-75 years
* Symptomatic limb weakness
* FSHD patients who use the wheelchair daily and are able to stand or to walk at most 30 meters with assistance, and wheelchair-bound patients who are unable to walk.
* Clinical severity score (CSS) ≥ 8
* Patient affiliated to the social security system
* Patient giving written consent after written and oral information.
* If taking over the counter supplements, willing to remain consistent with supplement regimen throughout the course of the study

Exclusion Criteria:

* Patients with comorbidity not related to the disease that can modify the natural evolution of the disease or would interfere with safe testing in the opinion of the Investigator
* Regular use of available muscle anabolic/catabolic agents such as corticosteroids, oral testosterone or derivatives, or oral beta agonists
* Use of an experimental drug in an FSHD clinical trial within the past 30 days
* Pregnancy
* Vulnerable person (person deprived of their administrative and legal liberty, hospitalized person for other purposes than research)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change of the Motor Function Measure-32 (MFM-32) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  Within MFM-32, 32 terms will be evaluated to describe patient's motor functions and grouped into 3 sub-scores at baseline, 6, 12 and 24 months:
  D1: standing position and transfer D2: axial and proximal motor function D3: distal motor function The MFM-32 ratings rely on the use of a 4-point Likert scale based on the subject's maximal abilities without assistance (0: cannot initiate the task or maintain the starting position; 1: performs the task partially; 2: performs the task incompletely or imperfectly; 3: performs the task fully and normally.)
Change of the Manual Muscle Testing (MMT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The Manual Muscle Testing is a modified Medical Research Council 13-point and is used with standardized positions for each grade and each muscle following the recommendations of the FSH-DY Group. Shoulder abduction and flexion, elbow flexion and extension, wrist flexion and extension, fingers flexion and extension, hip flexion and abd/adduction, knee flexion and extension, ankle plantarflexion and dorsiflexion strength will be measured bilaterally
Change of the Hand-Held dynamometry (HHD) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  Hand-Held dynamometry (HHD) assess the isometric muscle strength in both the upper and lower limbs bilaterally (global shoulder abduction and flexion, elbow flexion and extension, hip abduction, knee extension, ankle dorsiflexion isometric strength). The required equipment is a calibrated hand-held dynamometer (MicroFet). The patient has to push against the hand-held dynamometer 3 times as hard as he can for 3-5 seconds. The maximal value will be kept for further analysis.
Change of the Pinch and Grip test from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The purpose of those tests is to measure the maximum isometric strength of the hand and forearm muscles when doing a grasping or a pinching action. The equipment required for the grip and the pinch tests is a calibrate dynamometer. The subject should be strongly encouraged to give a maximum effort. We record three trials for each hand, alternating hands with at least 30 seconds recovery between each effort. We keep the best result.

SECONDARY OUTCOMES:
Change of the 9-Hole Peg test (9-HPT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The 9-Hole Peg Test is used to measure finger dexterity. The patient is seated at a table with a small, shallow container holding 9 pegs and a wood or plastic block containing nine empty holes. When a stopwatch is started, the patient picks up the 9 pegs one at a time as quickly as possible, puts them in the 9 holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to put the pegs and to remove them (one lap) will be recorded, 3 times alternating hands. The best trial will be registered for both hands.
Change of the repeated 9-Hole Peg test (r9-HPT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The repeated 9-Hole Peg test (r9-HPT) est a fatigability test. The same procedure like 9-HPT is repeated 5 times (5 laps) with the same hand. The total time to complete the r9-HPT is recorded and the ratio "last lap/first lap" is calculated. The patient will choose the tested hand.
Change of the classic Timed Up and Go test (classic TUG) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  Balance and mobility in patients able to walk at most 30 meters will be assessed using the classic Timed Up and Go test (TUG). The classic TUG measures, in seconds, the time taken by a patient to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm), walk 3 meters, turn, walk back to the chair, and sit down. The best performance will be recorded.
Change of the optimized Timed Up and Go test (classic TUG) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The optimized TUG test measures, in seconds, the time taken by patient to sit up from a lying down position (1st time interval); stand up from the mat (approximate height of 46 cm, walk 3 meters, turn, walk back to the mat, sit down (2nd time interval); and lie down to return to starting position (3rd time interval).
Change of the Sit Up test (SiUT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The SiUT measures, in seconds, the time taken by a patient to sit up from a lying down position and to return to the initial position.
Change of the repeated Sit Up test (r-SiUT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The r-SiUT measures, in seconds, the time taken by a patient to sit up from a lying down position and to return to the initial position (1 lap). This task is repeated 5 times (5 laps). The total time to complete the trial is recorded and the ratio last lap/first lap is calculated.
Change of the Stand Up test (SaUT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The SaUT measures, in seconds, the time taken by a patient to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm) and to return to the initial position.
Change of the repeated Stand Up test (r-SaUT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The r-SaUT measures, in seconds, the time taken by a patient to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm) and to return to the initial position. This task is repeated 5 times (5 laps). The total time to complete the trial is recorded and the ratio last lap/first lap is calculated.
Change of the Neck Flexion Fatigability Test (NFFT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The NFFT measures, in seconds, the total time that the patient can hold the following position: in a lying position, arm relaxed on each sides of the body, the patient has to raise his head from the table flexing his neck at 45°.
Change of the Bend Over Test (BOT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The BOT measures, in seconds, the time taken by the patient, to bend forward, knee in extension, to touch a support placed in front of the middle of the tibia and to return to the initial position.
Change of the repeated Bend Over Test (r-BOT) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The r-BOT measures, in seconds, the time taken by the patient, to perform 5 times consecutively the following task: to bend forward, knee in extension, to touch a support placed in front of the middle of the tibia and to return to the initial position.
Change of the muscle mass from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  Muscle mass is assessed with a portable device that quantify muscle volume and reconstruct the profile of muscle cross-sectional area along the thigh or leg. The device consists in a multifrequency bioelectrical impedance analyser, a pair of current electrodes, and a matrix of voltage electrodes positioned on the anterior thigh. Impedance will be measured on each thigh and each arm one after the other.
Change of the respiratory function (sitting and bedside spirometry) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  Sitting and bedside spirometry allow to obtain forced vital capacity and forced respiratory volume in 1 second, two standardized outcomes commonly used to evaluate respiratory function in clinical follow up and clinical trials.
Change of the Swallowing Quality of Life questionnaire (SWAL-QOL) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The original SWAL-QOL scale has 44 items exploring patient's quality of life and grouped into 10 lifestyle scales: burden of eating difficulty; eating duration; eating desire; food selection; communication; fear; mental health; social impact; fatigue; and sleep. There is also a symptom-frequency scale in which each item is scored from 1 to 5 (1 for poorest, 5 for best quality of life). For each scale, a separate score out of 100% is calculated, with each item having the same importance. There is no global score of QOL.
Change of the Sydney Swallow Questionnaire (SSQ) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The Sydney Swallow Questionnaire (SSQ) is a 17 question, self-report inventory, which was developed to measure symptomatic severity of oral-pharyngeal dysphagia as reported by the affected patient. The questionnaire uses a 100mm long visual analogue scale (VAS) for all but one question.
Change of the Fatigue Severity Scale (FSS) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The FSS is a unidimensional scale which focuses on the physical aspects of fatigue. It is a self-reported questionnaire developed to measure the impact of disabling fatigue on daily functioning. It covers several areas including physical, social, and cognitive effects. The FSS is a patient-reported outcome composed of 9-items with scores ranging from 1 = "strongly disagree" to 7 = "strongly agree".
Change of the Patient-Reported Outcomes Measurement Information System 57 (PROMIS57) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The PROMIS57 is an instrument developed by the NIH PROMIS initiative. The PROMIS®-57 scales include eight items from seven primary domains: depression, anxiety, physical function, pain interference (and pain intensity), fatigue, sleep disturbance, and satisfaction with social roles. A 5-point scale is used for each instrument, except for the 0-10 pain intensity item.
  Raw scores for each of the seven short forms (domains) in PROMIS-57 are calculated, and scores are converted to T-scores for each of the seven short forms (domains) in PROMIS-57 based on the PROMIS guidelines (http://www.healthmeasures.net).
  The T-score conversion establishes 50 as a general population mean for all PROMIS domains, and any 10-point deviation corresponds to one standard deviation (SD) difference, for easy-to-understand and consistent scoring across measures.
Change of the Upper Extremity Functional Index 15 (UEFI15) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The Upper Extremity Functional Index 15 (UEFI15) is a validated patient reported measure for adults with upper extremity dysfunction. This index measures upper extremity dysfunction. 20 questions are combined into a total score, the score is transformed into a normalized score with 80 representing normal, and lower scores representing increasing disability.
Change of the Facial Disability Index (FDI) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The Facial Disability Index (FDI) is a short 5 items questionnaire which assesses the physical impact of facial weakness. The five questions are summed into total score which transformed onto a percentage scale, with 100 representing normal, and lower scores representing increasing disability.
Change of the Multidimensional Dyspnea Profile (MDP) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The Multidimensional Dyspnea Profile (MDP) is a questionnaire which assesses overall breathing discomfort, sensory qualities, and emotional responses in laboratory and clinical settings. The MDP assesses dyspnea during a specific time or a particular activity (focus period) and is designed to examine individual items that are theoretically aligned with separate mechanisms.
Change of the Speech Handicap Index (SHI) from Baseline (T0) to 6 months (T6), 12 months (T12) and 24 months (M24) | at baseline, 6, 12 and 24 months
  The Speech Handicap Index (SHI) is one of the self-report assessments and questionnaires to assess speech problem and it is a test with 30 items.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided